# **Informed Consent Model for S1701**

This model informed consent form has been reviewed by the DCTD/NCI and is the official consent document for this study. Local IRB changes to this document are allowed. (Institutions should attempt to use sections of this document that are in bold type in their entirety.) Editorial changes to these sections may be made if they do not change information or intent. If the institutional IRB insists on making additions, deletions, or more substantive modifications to the risks or alternatives sections, they may be justified in writing by the investigator and approved by the IRB. Under these circumstances, the revised language, justification, and a copy of the IRB minutes must be forwarded to the SWOG Operations Office for approval before a patient may be registered to this study.

Please particularly note that the questions related to banking of specimens for future study are in bolded type and may not be changed in any way without prior approval from the SWOG Operations Office.

| Readability Statistics: | |
|----------------------------|---------------------------------|
| Flesch Reading Ease | <u>61.4</u> (targeted above 55) |
| Flesch-Kincaid Grade Level | 8.6 (targeted below 8.5) |

- Instructions and examples for informed consent authors are in [italics].
- A blank line, \_\_\_\_\_, indicates that the local investigator should provide the appropriate information before the document is reviewed with the prospective research participant.
- The term "study doctor" has been used throughout the model because the local investigator for a cancer treatment trial is a physician. If this model is used for a trial in which the local investigator is not a physician, another appropriate term should be used instead of "study doctor".
- The dates of protocol updates in the header and in the text of the consent is for reference to this model only and should not be included in the informed consent form given to the prospective research participant.
- The local informed consent must state which parties may inspect the research records. This includes the NCI, the drug manufacturer for investigational studies, any companies or grantors that are providing study support (these will be listed in the protocol's model informed consent form) and SWOG.
- "SWOG" must be listed as one of the parties that may inspect the research records in all protocol consent forms for which patient registration is being credited to SWOG. This includes consent forms for studies where all patients are registered directly through the SWOG Data Operations Office, all intergroup studies for which the registration is being credited to SWOG (whether the registration is through the SWOG Data Operations Office or directly through the other group), as well as



<sup>\*</sup>Notes for local institution informed consent authors:

- consent forms for studies where patients are registered via CTSU, and the registration is credited to SWOG.
- When changes to the protocol require revision of the informed consent document, the IRB should have a system that identifies the revised consent document, to preclude continued use of the older version and to identify file copies. An appropriate method to identify the current version of the consent is for the IRB to stamp the final copy of the consent document with the approval date. The stamped consent document is then photocopied for use. Other systems of identifying the current version of the consent such as adding a version or approval date are allowed if it is possible to determine during an audit that the patient signed the most current version of the consent form.

#### \*Notes for local investigators:

- The goal of the informed consent process is to provide people with sufficient information for making informed choices about participating in research. consent form provides a summary of the study, the individual's rights as a study participant, and documents their willingness to participate. The consent form is, however, only one piece of an ongoing exchange of information between the investigator and study participant. For more information about informed consent, review the "Recommendations for the Development of Informed Consent Documents for Cancer Clinical Trials" prepared by the Comprehensive Working Group on Informed Consent in Cancer Clinical Trials for the National Cancer Institute. The Web site address for this document http://cancer.gov/clinicaltrials/understanding/simplification-of-informed-consentdocs/
- Suggestion for Local Investigators: An NCI pamphlet explaining clinical trials is available for your patients. The pamphlet is titled: "Taking Part in Cancer Treatment Research Studies". This pamphlet may be ordered on the NCI Web site at <a href="https://cissecure.nci.nih.gov/ncipubs">https://cissecure.nci.nih.gov/ncipubs</a> or call 1-800-4- CANCER (1-800-422-6237) to request a free copy.
- Optional feature for Local Investigators: Reference and attach drug sheets, pharmaceutical information for the public, or other material on risks. Check with your local IRB regarding review of additional materials.



<sup>\*</sup>These notes for authors and investigators are instructional and should not be included in the informed consent form given to the prospective research participant.

# Study Title for Study Participants: Testing the Combination of Carboplatin – Paclitaxel with or Without Ramucirumab in Patients with Thymic Cancer

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>:

"S1701, A Randomized Phase II Trial of Carboplatin-Paclitaxel with or Without Ramucirumab in Patients with Unresectable Locally Advanced, Recurrent, or Metastatic Thymic Carcinoma"

## What is the usual approach to my thymic cancer?

You are being asked to take part in this study because you have thymic cancer which is not able to be treated with surgery. People who are not in a study are usually treated with radiation therapy, hormone therapy or chemotherapy with FDA approved drugs such as doxorubicin, epirubicin, cisplatin, carboplatin, cyclophosphamide, ifosfamide, vincristine, etoposide, paclitaxel, and pemetrexed.

## What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices. For example:

- you may choose to have the usual approach described above
- you may choose to take part in a different study if one is available
- you may choose not to be treated for cancer, but you may want to receive comfort care to relieve symptoms

# Who is doing this study?

SWOG is sponsoring this trial. SWOG is an adult cancer clinical trials organization. SWOG is funded through the National Cancer Institute, and its network consists of about four thousand physicians at almost three hundred institutions throughout the United States. Your study doctor has met all requirements to be a member of SWOG and to perform National Cancer Institute-funded research through this Group.

# Why is this study being done?

The purpose of this study is to compare any good and bad effects of using ramucirumab along with the usual chemotherapy combination (carboplatin and paclitaxel) to the usual chemotherapy combination alone. Ramucirumab is FDA-approved for non-small cell lung cancer but not for thymic cancer; however, ramucirumab in combination with carboplatin and paclitaxel is considered investigational and is not approved for this indication. Ramucirumab is a monoclonal antibody, a type of protein made in the laboratory that can bind to substances in the body, including cancer cells. Ramucirumab targets the vascular endothelial growth factor receptor 2 (VEGFR 2). VEGFR2 is an important molecule that supports the growth of blood vessels by a process called



angiogenesis. Growth of these blood vessels can feed tumors and cause them to grow. Ramucirumab blocks VEGFR2 and may prevent angiogenesis in advance thymic tumor patients. This study will allow the researchers to know whether this different approach is better, the same, or worse than the usual approach. To be better, the study approach should extend the amount of time you are cancer-free compared to the usual approach.

This chemotherapy combination, carboplatin, and paclitaxel has already been FDA-approved.

There will be about 66 patients taking part in this study.

## What are the study groups?

This study has 2 study groups.

- Group 1 will get carboplatin and paclitaxel with ramucirumab for 6 cycles. After 6 cycles of the carboplatin and paclitaxel with ramucirumab, you will receive ramucirumab alone on Day 1 of Cycle 7 and subsequent cycles for up to 1 year.
- Group 2 will get carboplatin and paclitaxel for 6 cycles.

The treatments on this study are described in the table below:

| Group | Drug | How often is it given? | How is it given? | What days is it given on? | What is the cycle duration? |
|---|---|---|---|---|---|
| 1 | Ramucirumab | Once, every 21 days, for up to one year | Into a vein, over 60 minutes | Day 1 | 21 days |
| 1 | Carboplatin | Once, every 21 days, cycles 1-6 | Into a vein | Day 1 | 21 days |
| 1 | Paclitaxel | Once, every 21 days, cycles 1-6 | Into a vein | Day 1 | 21 days |
| 2 | Carboplatin | Once, every 21 days cycles 1-6 | Into a vein | Day 1 | 21 days |
| 2 | Paclitaxel | Once, every 21 days cycles 1-6 | Into a vein | Day 1 | 21 days |

A computer will by chance assign you to treatment groups in the study. This is called randomization. This is done by chance because no one knows if one study group is better or worse than the other.

Another way to find out what will happen to you during this study is to read the chart below. Start reading at the left side and read across to the right, following the lines and arrows.





## How long will I be in this study?

You will receive the study treatment as long as the side effects are not too great and your disease does not get worse or until you have completed treatment. After you finish the study treatment, your doctor will continue to watch you for side effects and follow your condition for two years from the time you started the study.

## What extra tests and procedures will I have if I take part in this study?

All of the exams, tests, and procedures you will have are part of the usual approach for your cancer.

## What possible risks can I expect from taking part in this study?

#### If you choose to take part in this study, there is a risk that:

- You may lose time at work or home and spend more time in the hospital or doctor's office than usual
- You may be asked sensitive or private questions which you normally do not discuss
- The study drug(s)/study approach may not be better, and could possibly be worse, than the usual approach for your cancer.

The drugs used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will be testing your blood and will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the study drugs.

#### Here are important points about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.
- Some side effects may interfere with your ability to have children.
- Some side effects may be serious and may even result in death.



# Here are important points about how you and the study doctor can make side effects less of a problem:

- Tell the study doctor if you notice or feel anything different so they can see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce side effects.

The tables below show the most common and the most serious side effects that researchers know about. There might be other side effects that researchers do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

#### **Possible Side Effects of Carboplatin**

#### Common, some may be serious

In 100 people receiving carboplatin, more than 20 and up to 100 may have:

- Hair loss
- Vomiting, nausea
- Infection, especially when white blood cell count is low
- Anemia which may cause tiredness, or may require blood transfusions
- Bruising, bleeding
- Belly pain

#### Occasional, some may be serious

In 100 people receiving carboplatin, from 4 to 20 may have:

- Diarrhea, Constipation
- Numbness and tingling in fingers and toes
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Changes in taste
- Changes in vision

#### Rare, and serious

In 100 people receiving carboplatin, 3 or fewer may have:

• Damage to organs which may cause hearing and balance problems



#### **Possible Side Effects of Paclitaxel**

#### Common, some may be serious

In 100 people receiving paclitaxel, more than 20 and up to 100 may have:

- Anemia which may cause tiredness, or may require blood transfusions
- Infection, especially when white blood cell count is low
- Diarrhea, nausea, vomiting
- Sores in mouth which may cause difficulty swallowing
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Bruising, bleeding
- Pain
- Muscle weakness
- Numbness, tingling or pain of the arms and legs
- Hair loss

#### Occasional, some may be serious

In 100 people receiving paclitaxel, from 4 to 20 may have:

- Abnormal heartbeat
- Damage to the lungs which may cause shortness of breath
- Blood clot which may cause swelling, pain, shortness of breath

#### Rare, and serious

In 100 people receiving paclitaxel, 3 or fewer may have:

- Heart attack or heart failure which may cause shortness of breath, swelling of ankles, and tiredness
- A tear or a hole in the stomach which may cause belly pain or that may require surgery



## **Group 1 only**

#### Possible Side Effects of Ramucirumab

(Table Version Date: April 2022)

## Common, some may be serious

In 100 people receiving ramucirumab, more than 20 and up to 100 may have:

• Pain in belly

#### Occasional, some may be serious

In 100 people receiving ramucirumab, from 4 to 20 may have:

- Anemia which may cause tiredness, or may require blood transfusion
- An infection due to low white blood cells that may include fever, pain, redness, and/or difficulty breathing
- High blood pressure
- Diarrhea
- Headache
- Nosebleed
- Rash



#### Rare, and serious

In 100 people receiving ramucirumab, 3 or fewer may have:

- Heart failure (heart stops beating) which may cause shortness of breath, chest pain, swelling
  of ankles, and tiredness
- Stroke which may cause paralysis, weakness, or headache
- Blockage of the bowels which may cause pain, or vomiting
- A tear or hole in the stomach and/or bowel which may cause pain and may require surgery

Ramucirumab side effects have been observed in other clinical trials such as:

- Bleeding in the belly,
- Infusion related reaction which may cause fever, chills, rash, low blood pressure,
- Abnormal healing,
- Brain damage (possible headache, confusion, seizures, and/or vision loss), and kidney damage which may cause swelling, and may require dialysis.

Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

**Reproductive risks:** You should not get pregnant, breastfeed, or father a baby while in this study. The drugs used in this study could be very damaging to an unborn baby. Continue to use approved forms of birth control while receiving treatment, and for 4 months after the last dose of study drug. Check with the study doctor about what types of birth control, or pregnancy prevention, to use while in this study.

# What possible benefits can I expect from taking part in this study?

It is not possible to know at this time if the study drug(s)/study approach is better than the usual approach so this study may or may not help you. This study will help researchers learn things that will help people in the future.

# Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let the study doctor continue to provide your medical information to the organization running the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If new information becomes available
- If you do not follow the study rules



• If the study is stopped by the sponsor, IRB or FDA.

## What are my rights in this study?

Taking part in this study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not lose medical care or any legal rights.

## What are the costs of taking part in this study?

If you are selected for the group that will receive ramucirumab, the ramucirumab will be supplied at no charge while you take part in this study. The cost of getting the ramucirumab ready and giving it to you is not paid by the study sponsor so you or your insurance company may have to pay for this. It is possible that the ramucirumab may not continue to be supplied while you are on the study. Although not likely, if this occurs, your study doctor will talk to you about your options.

You and/or your health plan/insurance company will need to pay for the cost of carboplatin and paclitaxel; this will include the cost of getting carboplatin and paclitaxel ready and giving it to you. You and/or your health plan/insurance company will need to pay for all of the other costs of treating your cancer while in this study, including the cost of tests, procedures, or medicines to manage any side effects, unless you are told that certain tests are supplied at no charge. Before you decide to be in the study, you should check with your health plan or insurance company to find out exactly what they will pay for.

You will **not** be paid for taking part in this study.

# What happens if I am injured or hurt because I took part in this study?

If you are injured or hurt as a result of taking part in this study and need medical treatment, please tell your study doctor. The study sponsors will not offer to pay for medical treatment for injury. Your insurance company may not be willing to pay for study-related injury. If you have no insurance, you would be responsible for any costs.

If you feel this injury was a result of medical error, you keep all your legal rights to receive payment for this even though you are in a study.



## Who will see my medical information?

Your privacy is very important to us and the researchers will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you. Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database.

There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- The study sponsor and any drug company supporting the study, SWOG, Eli Lilly and Company, and Bristol Myers Squibb.
- The Institutional Review Board, IRB, is a group of people who review the research with the goal of protecting the people who take part in the study.
- The Food and Drug Administration and the National Cancer Institute in the U.S., and similar ones if other countries are involved in the study.

## Where can I get more information?

You may visit the NCI Web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this website at any time.

# Who can answer my questions about this study?

| You can talk to the stud | ly doctor about any questions or concerns | you have about this study or to |
|---|---|---|
| report side effects or inju | uries. Contact the study doctor | (insert name of study |
| doctor[s]) at | (insert telephone number). | |



#### Additional studies section:

This section is about optional studies you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. You will not get health benefits from any of these studies. The researchers leading this optional study hope the results will help other people with cancer in the future.

The results will not be added to your medical records and you or your study doctor will not know the results.

You will not be billed for these optional studies. You can still take part in the main study even if you say 'no' to any or all of these studies. If you sign up for but cannot complete any of the studies for any reason, you can still take part in the main study.

Circle your choice of "yes" or "no" for the following:

#### **Future Contact**

I agree to allow my study doctor, or someone approved by my study doctor, to contact me regarding future research involving my participation in this study.

Yes No

# **Optional Sample Collections for Biobanking for Possible Future Studies**

Researchers are trying to learn more about cancer, diabetes, and other health problems. Much of this research is done using samples from your tissue, blood, urine, or other fluids. Through these studies, researchers hope to find new ways to prevent, detect, treat, or cure health problems.

Some of these studies may be about genes. Genes carry information about features that are found in you and in people who are related to you. Researchers are interested in the way that genes affect how your body responds to treatment.

If you choose to take part, a sample of tissue from your previous biopsy and a blood sample will be collected. The researchers ask your permission to store and use your samples and related health information (for example, your response to cancer treatment, results of study tests and medicines you are given) for medical research. The research that may be done is unknown at this time. Storing samples for future studies is called "biobanking". The Biobank is being run by SWOG and supported by the National Cancer Institute.



#### What is involved?

If you agree to take part, here is what will happen next:

- 1) About ½ a tablespoon of blood will be collected from a vein in your arm at 3 timepoints during the study (pre-study, Cycle 3, end of study treatment).
- 2) A sample from the tissue that was collected at the time of your surgery will be sent to the Biobank.
- 3) Your sample and some related health information may be stored in the Biobank, along with samples and information from other people who take part. The samples will be kept until they are used up. Information from your medical record will be updated from time to time.
- 4) Qualified researchers can submit a request to use the materials stored in the Biobanks. A science committee at the clinical trials organization, and/or the National Cancer Institute, will review each request. There will also be an ethics review to ensure that the request is necessary and proper. Researchers will not be given your name or any other information that could directly identify you.
- 5) Neither you nor your study doctor will be notified when research will be conducted or given reports or other information about any research that is done using your samples.
- 6) Some of your genetic and health information may be placed in central databases that may be public, along with information from many other people. Information that could directly identify you will not be included.

## What are the possible risks?

- 1) The most common risks related to drawing blood from your arm are brief pain and possibly a bruise.
- 2) There is a risk that someone could get access to the personal information in your medical records or other information researchers have stored about you.
- 3) There is a risk that someone could trace the information in a central database back to you. Even without your name or other identifiers, your genetic information is unique to you. The researchers believe the chance that someone will identify you is very small, but the risk may change in the future as people come up with new ways of tracing information.
- 4) In some cases, this information could be used to make it harder for you to get or keep a job or insurance. There are laws against the misuse of genetic information, but they may not give full protection. There can also be a risk in knowing genetic information. New health information about inherited traits that might affect you or your blood relatives could be found during a study. The researchers believe the chance these things will happen is very small, but cannot promise that they will not occur.



## How will information about me be kept private?

Your privacy is very important to the researchers, and they will make every effort to protect it. Here are just a few of the steps they will take:

- 1) When your sample(s) is sent to the researchers, no information identifying you (such as your name) will be sent. Samples will be identified by a unique code only.
- 2) The list that links the unique code to your name will be kept separate from your sample and health information. Any Biobank and SWOG staff with access to the list must sign an agreement to keep your identity confidential.
- 3) Researchers to whom SWOG sends your sample and information will not know who you are. They must also sign an agreement that they will not try to find out who you are.
- 4) Information that identifies you will not be given to anyone, unless required by law.
- 5) If research results are published, your name and other personal information will not be used.

## What are the possible benefits?

You will not benefit from taking part. The researchers, using the samples from you and others, might make discoveries that could help people in the future.

## Are there any costs or payments?

There are no costs to you or your insurance. You will not be paid for taking part. If any of the research leads to new tests, drugs, or other commercial products, you will not share in any profits.

| What if I change m | y mind? | |
|---|---|---|
| • | longer want your samples to be used, ynsert name of study doctor for main trial) a | |
| any sample that remains | or of study doctor for main trial) who will in the bank will no longer be used and related information that have alreturned. | lated health information will no |
| What if I have mor | e questions? | |
| You can talk to the stud | y doctor about any questions or concerns | you have about this study or to |
| report side effects or inju | ries. Contact the study doctor | (insert name of study |
| doctor[s]) at | (insert telephone number). | <u> </u> |
| Please circle your answe | er to show whether you would like to take | part in each option: |
| Samples for futur | re research studies | |

My samples and related information may be kept in a Biobank for use in future health

This is the end of the section about optional studies.

NO

research.

YES



# My Signature Agreeing to Take Part in the Main Study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed copy of this form. I agree to take part in the main study.

| Participant's signature | <br> |
|-------------------------|------|
| Date of signature | |



## **Specimen Consent Supplemental Sheets**

## **How are Specimens Used for Research?**

#### Where do specimens come from?

A specimen may be from a blood sample or from bone marrow, skin, toenails, or other body materials. People who are trained to handle specimens and protect donors' rights make sure that the highest standards of quality control are followed by SWOG. Your doctor does not work for SWOG but has agreed to help collect specimens from many patients. Many doctors across the country are helping in the same way.

#### Why do people do research with specimens?

Research with specimens can help to find out more about what causes cancer, how to prevent it, how to treat it, and how to cure it. Research using specimens can also answer other health questions. Some of these include finding the causes of diabetes and heart disease or finding genetic links to Alzheimer's.

## What type of research will be done with my specimen?

Many kinds of studies use specimens. Some researchers may develop new tests to find diseases. Others may develop new ways to treat or even cure diseases. In the future, some of the research may help to develop new products, such as tests and drugs. Some research looks at diseases that are passed on in families (called genetic research). Research done with your specimen may look for genetic causes and signs of disease.

## How do researchers get the specimen?

Researchers from universities, hospitals, and other health organizations conduct research using specimens. They contact SWOG and request samples for their studies. SWOG reviews the way that these studies will be done and decides if any of the samples can be used. SWOG gets the specimen and information about you from your hospital and sends the specimen samples and some information about you to the researcher. SWOG will not send your name, address, phone number, social security number or any other identifying information to the researcher.

# Will I find out the results of the research using my specimen?

You will not receive the results of research done with your specimen. This is because research can take a long time and must use specimen samples from many people before results are known. Results from research using your specimen may not be ready for many years and will not affect your care right now, but they may be helpful to people like you in the future.

# Why do you need information from my health records?

To do research with your specimen, researchers may need to know some things about you. (For example: Are you male or female? What is your race or ethnic group? How old are you? Have you ever smoked?) This helps researchers answer questions about diseases. The information that will be given to the researcher may include your age, sex, race, diagnosis, treatments, and family history. This information is collected by your hospital from your health record and sent to SWOG. If more information is needed, SWOG will send it to the researcher.



## Will my name be attached to the records that are given to the researcher?

No. Your name, address, phone number and anything else that could identify you will be removed before they go to the researcher. The researcher will not know who you are.

## How could the records be used in ways that might be harmful to me?

If your confidential genetic information is discovered, you may suffer from genetic discrimination. Genetic discrimination occurs if people are treated unfairly because of differences in their genes that increase their chances of getting a certain disease. In the past, this could have resulted in the loss of health insurance or employment. Because of this, The Genetic Information Nondiscrimination Act of 2008, also referred to as GINA, was passed by Congress to protect Americans from such discrimination. The new law prevents discrimination from health insurers and employers. This act was signed into federal law on May 21, 2008, and went into effect May 2009. This law does not cover life insurance, disability insurance and long-term care insurance.

While this study has safeguards in place to protect your confidential genetic information and to make it extremely unlikely that your identity would be connected with any special studies that are performed on your tissue, it is possible that this information could be discovered by someone who is unauthorized to have access to it.

#### **How am I protected?**

SWOG oversees making sure that information about you is kept private. SWOG will take careful steps to prevent misuse of records. Your name, address, phone number and any other identifying information will be taken off anything associated with your specimen before it is given to the researcher. This would make it very difficult for any research results to be linked to you or your family. Also, people outside the research process will not have access to results about any one person which will help to protect your privacy.

## What if I have more questions?

If you have any questions, please talk to your doctor, or nurse, or call our research review board at (Insert IRB's Phone Number).

